CLINICAL TRIAL: NCT00215345
Title: A Phase II Trial of Combination Therapy With Celecoxib and Taxotere for the Treatment of Stage D3 Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Veterans Affairs, New Jersey (U.S. Federal Agency)
Collaborators: Pfizer (Industry); Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COXAON-0509-047; GIA16125
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Prostate Cancer
Keywords: Celecoxib; Taxotere; Hormone Refractory Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Celecoxib

INTERVENTIONS:
Drug: Taxotere
Drug: Celecoxib

SUMMARY:
The purpose of this clinical trial is to find out the safety and effectiveness as well as patient's quality of life on the combination of Taxotere and celecoxib on patients with hormone refractory prostate cancer. Celecoxib (Celebrex) is an FDA approved drug to treat arthritis. Taxotere (Docetaxel) is an FDA approved chemotherapy drug to treat certain forms of cancer. Both drugs have demonstrated evidences of tumor blood vessel suppression and combination of these two drugs could possibly arrest further tumor growth or make the tumor decrease in size.

DETAILED DESCRIPTION:
The standard hormone therapy for patients with metastases is androgen deprivation. This treatment leads to response in 75-80% of the patients, with median duration of response of only 14-18 months. Once the patient becomes hormone resistant, there is no effective therapy to prolong life. For patients with HRPC, the median life expectancy is 17 months.2 Thus palliative care remains the standard therapy for HRPC. The most widely used chemotherapy regimens are combinations of mitoxantrone with prednisone and taxanes with estramustine phosphate.3,4,5 Taxotere has also demonstrated activity in prostate cancer cell lines.6 Several clinical studies have demonstrated its activity in patients with metastatic prostate cancer as a single agent or in combination.4, 5 Taxotere may exert its effects in part through anti-angiogenic effects.7 Recent work in animal models has provided additional evidence for the beneficial role of angiostatic agents in the treatment of malignant diseases. This is the first study of the two drugs used together in prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically proven adenocarcinoma of the prostate gland.
* Patient must have evidence of progressive metastatic disease (e.g., bone, pelvic mass, lymph node, liver or lung metastases) within 6 weeks prior to participation in the study.
* Patients who have evaluable but not measurable disease must not have an elevated PSA level as the only evidence of disease. While castrated, the patients should have rising PSA on two consecutive measurements at least 1 week apart. The confirmatory PSA must be obtained within 1 week prior to study registration and should be >10ng/ml.
* Patients with bone metastases only (i.e., lacking soft-tissue disease) must have a PSA level of > 10 ng/ml. Patients with soft tissue metastases and /or visceral disease must have either measurable disease or a PSA level of > 10 ng/ml.
* Radiological evidence of hydronephrosis will not by itself constitute evidence of metastatic disease.
* Patients must have had prior treatment with bilateral orchiectomy or other primary hormonal therapy (e.g., estrogen therapy, LHRH analog + flutamide, etc.) with evidence of treatment failure.

NOTE: patients who have not undergone bilateral orchiectomy must continue LHRH agonist therapy (e.g., depot leuprolide or goserelin) while receiving this protocol therapy. For these patients the testosterone level should be preferably checked before enrollment and should be < 50 ng/dl.

* For patients previously treated with flutamide (Eulexin), nilutamide (Nilandron), or bicalutamide (Casodex): Patients must have discontinued flutamide or nilutamide < 4 weeks and for bicalutamide 6 weeks prior to registration.
* Patients must not have received prior treatment with chemotherapy within the last 5 years.
* Patients must not have had prior radiotherapy < 4 weeks prior to this protocol treatment.
* Patients must not have previously received Strontium 89, Samarium 153, or other radioisotope therapies.
* Patients must have recovered from all toxicities due to prior treatment for prostate cancer prior to receiving this protocol treatment.
* Patients must have adequate bone marrow function: (WBC > 4000/ mm3, granulocytes > 1500/ mm3, platelet count > 100,000/mm3, and Hemoglobin > 8.0 g/dl < 4 weeks prior to participate in this study.
* Patients must have the following chemistry values < 4 weeks prior to participate in this study:
* Total bilirubin must be within normal limits.
* Creatinine < 2.0 mg/d. or creatinine clearance > 50 ml/min
* Transaminases (SGOT and/or SGPT) may be up to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphastase is < ULN, or alkaline phosphastase may be up to 4 x ULN if transaminases are < ULN.
* Peripheral neuropathy must be < grade 1
* Patients must have no active angina pectoris, or known heart disease of New York Heart Association Class III-IV. Patients must not have a history of myocardial infarction < 6 months prior to the study participation.
* Patients with a history of prior malignancy are eligible provided they were treated with curative intent and have been free of disease for the time period considered appropriate for the specific cancer.
* No serious concurrent medical illness or active infection should be present which would jeopardize the ability of the patient to receive the chemotherapy outlined in this protocol with reasonable safety.
* Sexually active patients must use an accepted and effective method of contraception while receiving protocol treatment.
* Patients must have a Karnofsky Performance Scale (KPS) score over 50. (equaling ECOG Performance Scale of 0, 1, or 2).
* Age > 18 years

Exclusion Criteria:

* Patients with a history of severe hypersensitivity to Taxotere or other drugs formulated with polysorbate 80 must be excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2002-08; Study Completion 2006-12

PRIMARY OUTCOMES:
Determine the effect of Taxotere and celecoxib on PSA and objective response in patients with HRPC

SECONDARY OUTCOMES:
Evaluate the toxicity of the combination of celecoxib and Taxotere in patients with stage D3 prostate cancer.
Determine the effects of this regimen on quality of life.
Determine the survival of the patients treated

CONTACTS AND LOCATIONS:
Overall Officials: Basil Kasimis, MD, Principal Investigator — Department of Veterans Affairs NJ Health Care System
Locations (1):
- Department Of Veterans Affairs NJ Health Care System, East Orange, New Jersey, United States

REFERENCES:
- [Result] Kasimis B, Cogswell J, Hwang S, Chang VT, Srinivas S, Zhong F, Duque L, Morales E, Boholli I, Blumenfrucht M: High Dose Celecoxib © and Docetaxel (D) in Patients (pts) with Hormone Resistant Prostate Cancer (HRPC). Results of an Ongoing Phase II Trial Proc Am Soc Clin Oncol, Vol 24#4704, 2005
- [Result] Yudd M, Kasimis B, Hwang S, Stanislaus G, Mcdowall S, Haastrup A, Penix J, Boholli I, Xia Q, Nazha N: Renal Effects of High Dose Celecoxib © during 2 Phase II Trials for Hormone Resistant Prostate Cancer (HRPC) Proc Am Soc Clin Oncol, Vol 24# 4751, 2005.